CLINICAL TRIAL: NCT04408846
Title: An Open-Label Randomized Controlled Study of the Efficacy of Surgical Treatment in Patients With Single Level Lumbar Spinal Stenosis Using Minimally Invasive Surgery and Traditional Open Surgical Procedure
Brief Title: Minimally Invasive Surgery Versus Traditional Open Surgery In The Treatment Of Single Level Lumbar Stenosis
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The Study will be conducted in another research center. The Sponsor has changed.
Sponsor: Novosibirsk Research Institute of Traumatology and Orthopaedics n.a. Ya.L. Tsivyan (Other Government)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: NS02-01
Record Dates: First submitted 2020-05-20; First posted 2020-05-29 (Actual); Last update posted 2020-09-11 (Actual); Status verified 2020-05

CONDITIONS: Intervertebral Disc Degeneration; Lumbar Spinal Stenosis
MeSH Terms: conditions — Intervertebral Disc Degeneration; Spinal Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Minimally invasive lumbar fusion (Other)
  Interventions: Device: Lumbar fusion
- Open posterior lumbar fusion (Other)
  Interventions: Device: Lumbar fusion

INTERVENTIONS:
Device: Lumbar fusion — Patients will receive a single level instrumented fusion using a minimally invasive or open traditional surgical procedure with a posterior fixation. For the use of a posterior fixation system, the CD Horizon® Spinal System, is mandatory in this study and will be either minimally invasive or open.

SUMMARY:
The purpose of this study is to determine the effectiveness of minimally invasive surgical technique over the traditional open surgical procedure in patients with degenerative lumbar stenosis

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 75 years;
* Patient has single level degenerative lumbar spinal stenosis and an indication for a single level instrumented lumbar fusion for the treatment;
* Symptoms persisting for at least three months prior to surgery;
* Given written Informed Consent;
* Able and agree to fully comply with the clinical protocol and willing to adhere to follow-up schedule and requirements.

Exclusion Criteria:

* Prior lumbar spinal fusion at any level;
* Other non-degenerative spinal conditions (e.g. infectious, traumatic, metabolic, inflammatory, neoplastic, structural or other pathology) that may have an impact on subject safety, wellbeing or the intent and conduct of the study;
* Any condition that cannot be treated with mini-invasive unilateral decompression and fusion;
* History or presence of any other major neurological disease or condition that may interfere with the study assessments (e.g. significant peripheral neuropathy, multiply sclerosis);
* Previous enrollment in this study, current enrollment or plans to be enrolled in another study (in parallel to this study).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-12-01 (Estimated); Primary Completion 2021-12-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Oswestry Disability Index (ODI) | 3 months
  To observe the change of ODI as compared to baseline through follow-up terms

SECONDARY OUTCOMES:
Change from baseline in Oswestry Disability Index (ODI) | Through 2 years
  To observe the change of ODI as compared to baseline through follow-up terms
Change from baseline in Numeric Pain Rating Score (NPRS) | Through 2 years
  To observe the change of NPRS as compared to baseline through follow-up terms
Change from baseline in EuroQol Five-Dimensional descriptive system questionnaire (EQ-5D) | Through 2 years
  To observe the change of EQ-5D as compared to baseline through follow-up terms
Change from baseline in Douleur Neuropathique 4 (DN4) | Through 2 years
  To observe the change of DN4 as compared to baseline through follow-up terms
Change from baseline in The Health Transition Item from SF-36 (HTI Item) | Through 2 years
  To observe the change of HTI Item through follow-up terms
Change from baseline in Clinical Global Impression Of Change (CGIC) scale | Through 2 years
  To observe the change of CGIC through follow-up terms
Fusion rate success | 12 months and 24 months post op
  Interbody fusion rate on CT based on Tan grades
Cost-effectiveness | 14th day of hospital stay
  Total cost of surgical procedure (implanted system, the salary for surgery team) and the cost of patient's staying at the clinic before discharge.
Adverse Events | Through 2 years
  Document Adverse Events (incl. adverse events related to device) occurrence throughout the study

CONTACTS AND LOCATIONS:
Locations (1):
- Novosibirsk Research Institute of Traumatology and Orthopaedics n.a. Ya.L. Tsivyan, Novosibirsk, Russia